CLINICAL TRIAL: NCT05484206
Title: A Phase 1 Open-Label, Single-Dose, Parallel-Group Study of the Pharmacokinetics and Safety of VIR-2218 and VIR-3434 Monotherapy and Combination Therapy in Adult Participants With Hepatic Impairment
Brief Title: Effect of Hepatic Impairment on the Pharmacokinetics and Safety of VIR-2218 and VIR-3434
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-2218-V107
Record Dates: First submitted 2022-07-15; First posted 2022-08-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Impairment; Cirrhosis
Keywords: siRNA; Monoclonal antibody; HDV; Compensated Cirrhosis; Decompensated Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: CPT-B (moderate HI) participants and matched healthy participants will be evaluated first (Experimental): All participants in Cohort 1 will be receiving VIR-2218 monotherapy.
  Interventions: Drug: VIR-2218
- Cohort 2: CPT-C (severe HI) participants and matched healthy participants (Experimental): This arm is optional based on Cohort 1. All participants in Cohort 2 will be receiving VIR-2218 monotherapy.
  Interventions: Drug: VIR-2218
- Cohort 3: CPT-A (mild HI) participants and matched healthy participants (Experimental): This cohort is optional. All participants in Cohort 3 will be receiving VIR-2218 monotherapy.
  Interventions: Drug: VIR-2218
- Cohort 4: CPT-A (mild HI) participants and matched healthy participants (Experimental): All participants in Cohort 4 will be receiving VIR-3434 monotherapy.
  Interventions: Drug: VIR-3434
- Cohort 5: CPT-B (moderate HI) participants and matched healthy participants (Experimental): All participants in Cohort 5 will be receiving VIR-3434 monotherapy.
  Interventions: Drug: VIR-3434
- Cohort 6: CPT-C (severe HI) participants and matched healthy participants (Experimental): This arm is optional based on Cohort 5. All participants in Cohort 6 will be receiving VIR-3434 monotherapy.
  Interventions: Drug: VIR-3434
- Cohort 7: CPT-A (mild HI) and matched healthy participants (Experimental): All participants in Cohort 7 will be receiving VIR-3434 and VIR-2218 combination therapy.
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 8: CPT-B (moderate HI) and matched healthy participants (Experimental): All participants in Cohort 8 will be receiving VIR-3434 and VIR-2218 combination therapy.
  Interventions: Drug: VIR-2218; Drug: VIR-3434
- Cohort 9: CPT-C (severe HI) and matched healthy participants (Experimental): This arm is optional based on Cohort 8. All participants in Cohort 9 will be receiving VIR-3434 and VIR-2218 combination therapy.
  Interventions: Drug: VIR-2218; Drug: VIR-3434

INTERVENTIONS:
Drug: VIR-2218 — VIR-2218 given by subcutaneous injection.
  Arms: Cohort 1: CPT-B (moderate HI) participants and matched healthy participants will be evaluated first; Cohort 2: CPT-C (severe HI) participants and matched healthy participants; Cohort 3: CPT-A (mild HI) participants and matched healthy participants; Cohort 7: CPT-A (mild HI) and matched healthy participants; Cohort 8: CPT-B (moderate HI) and matched healthy participants; Cohort 9: CPT-C (severe HI) and matched healthy participants
Drug: VIR-3434 — VIR-3434 given by subcutaneous injection.
  Arms: Cohort 4: CPT-A (mild HI) participants and matched healthy participants; Cohort 5: CPT-B (moderate HI) participants and matched healthy participants; Cohort 6: CPT-C (severe HI) participants and matched healthy participants; Cohort 7: CPT-A (mild HI) and matched healthy participants; Cohort 8: CPT-B (moderate HI) and matched healthy participants; Cohort 9: CPT-C (severe HI) and matched healthy participants

SUMMARY:
In this study, a single dose of VIR-2218 up to 200 mg SC or VIR-3434 at 300 mg SC monotherapy or a combination of VIR-2218 and VIR-3434 will be administered to assess the pharmacokinetic (PK) exposure, safety, and tolerability of VIR-2218 and VIR-3434 in participants with cirrhosis and Hepatic Impairment, defined using the Child-Pugh-Turcotte (CPT) categorization.

DETAILED DESCRIPTION:
Participants may be enrolled in Cohorts 1, 2, 3, 4, 5, 6, 7, 8, and 9 in a non-randomized way.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18 to ≤70 years of age at screening
* Must have a calculated BMI from 18.5 ≤ BMI ≤ 40 kg/m2
* All participants must have an eGFR ≥ 60 mL/min as calculated by the Modification of Diet in Renal Disease (MDRD) equation

Inclusion criteria: Healthy matched participants

* Must in the opinion of the Investigator, be in good health based upon medical history, vital signs, physical examination, and screening laboratory evaluations

Inclusion criteria: Hepatic impaired participants

* Apart from hepatic insufficiency, participants must, in the opinion of the Investigator be sufficiently healthy for study participation based on medical history, physical examination, vital signs, and screening laboratory evaluations
* Participant is considered to have chronic, stable moderate, severe, mild HI (of any etiology excluding chronic HBV and HDV) and has been clinically stable per Investigator assessment for at least 1 month prior to screening
* CPT score of 5 to 6 for mild HI at screening
* CPT score 7-9 for moderate HI at screening
* CPT score 10-15 severe HI at screening

Exclusion Criteria:

* Participants with unstable cardiac function or evidence of previous myocardial infarction in the past 12 months or any clinically significant active cardiovascular disease that, in the opinion of the Investigator, could interfere with the safety of the participant
* Any clinically significant conduction abnormality or arrhythmia (including non-sustained or sustained ventricular tachycardia as per Investigator's assessment)
* Infection with human immunodeficiency virus (HIV), hepatitis A virus (HAV), HBV (positive HBsAg or positive hepatitis B core antibody with negative hepatitis B surface antibody), hepatitis C virus (HCV), HDV or hepatitis E virus (HEV). HCV antibody positive participants with a negative HCV RNA are eligible. HDV antibody positive participants with a negative HDV RNA are eligible

Exclusion criteria: Healthy matched participants

* Systolic BP is outside the range of 90-160 mmHg, or diastolic BP is outside the range of 45-95 mmHg or heart rate is outside the range of 50-100 beats per minute (bpm) for female participants or 45-100 bpm for male participants at screening
* Use of any prescription medications or over-the-counter medications (with the exception of vitamins and/or hormonal contraceptive medication) within 30 days prior to D1 of study participation

Exclusion criteria: Participants with Hepatic impairment

* Not on stable dose and regimen of any medication
* Acute or worsening chronic hepatitis
* Participants requiring paracentesis more than once a month
* Participants with refractory encephalopathy or significant Central Nervous System
* History of gastric or esophageal variceal bleeding within the past 6 months
* Participants with Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement
* Presence of hepatopulmonary or hepatorenal syndrome
* Presence of primarily cholestatic liver diseases
* History of or currently listed for liver transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum observed Plasma concentration (Cmax) of VIR-2218 and metabolite AS(N-1)3'VIR2218 | 5 days
Area Under The Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUClast) of VIR-2218 and metabolite AS(N-1)3'VIR2218 | 5 days
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of VIR-2218 metabolite AS(N-1)3'VIR2218 | 5 days
Maximum observed Plasma concentration (Cmax) of VIR-3434 | 18 weeks
Area Under The Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUClast) of VIR-3434 | 18 weeks
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of VIR-3434 | 18 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to 18 Weeks
Incidence of ADA and titers of ADA to VIR-3434 at each study visit for cohorts receiving VIR-3434 therapy | 18 Weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Inland Empire Clinical Trials, Rialto, California
  - Orange County Research Center, Tustin, California
  - CenExel Research Centers of America, Hollywood, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Texas Liver Institute, San Antonio, Texas